CLINICAL TRIAL: NCT01082302
Title: An Open-Label, Single-Center Phase I (Phase IV/ USA) Study to Assess the Pharmacokinetic Profile of Topically Applied Veregen® 15% in Patients With External Genital and Perianal Warts Compared With Oral Intake of a Green Tea Beverage
Brief Title: Pharmacokinetic Study of Topically Applied Veregen 15% Compared With Oral Intake of Green Tea Beverage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MediGene (Industry)
Collaborators: Charité Research Organisation GmbH (Other)
Responsible Party: Dr. Petra Weyrauch, MediGene
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 1022; 2007-005432-88 (EudraCT Number)
Record Dates: First submitted 2010-02-01; First posted 2010-03-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Genital Warts; Perianal Warts
Keywords: green tea extract; Polyphenon E; Pharmacokinetics
MeSH Terms: conditions — Condylomata Acuminata | interventions — polyphenon E; green tea extract polyphenone E; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral intake of green tea beverage (Active Comparator): Healthy volunteers are asked to drink a defined amount of green tea beverage over 7 days
  Interventions: Other: Green Tea Beverage with defined catechin content
- Polyphenon E 15% ointment (Experimental): 3 times daily application of Polyphenon E 15% ointment on genital and perianal warts over 7 days
  Interventions: Drug: Polyphenon E (Veregen) 15% ointment

INTERVENTIONS:
Drug: Polyphenon E (Veregen) 15% ointment — 3 times daily application on genital and perianal warts over 7 days
  Arms: Polyphenon E 15% ointment
Other: Green Tea Beverage with defined catechin content — 3 times daily oral intake over 7 days
  Arms: oral intake of green tea beverage

SUMMARY:
This open, monocentric study is designed to investigate plasma concentrations of certain catechins after topical application of Veregen 15% ointment to genital or perianal warts in comparison to catechin plasma concentrations after oral intake of a defined dose of green tea beverage. The study is intended to demonstrate that topical administration of Veregen 15% induces catechin plasma concentrations lower or equivalent to those that can be reached with normal consumption of green tea.

ELIGIBILITY:
Inclusion Criteria:

For both subject groups (treatment arms 1 + 2):

1. Male and female subjects, 18 years of age or older at the time of enrollment. Subjects will be stratified by gender.
2. Written informed consent.
3. Ability to comply with the requirements of the study.

   For patients (treatment arm 1, additionally):
4. Clinical diagnosis of external genital and perianal warts which can be located: in men: over the glans penis, foreskin, penis shaft, and scrotum; in women: on the vulva; in both gender: in the inguinal, perineal, and perianal areas.
5. A total wart area of at least 100 mm² and a maximum of 2500 mm².
6. For women of child-bearing potential: negative pregnancy test and willingness to use two effective methods of contraception throughout their study participation is mandatory (oral contraceptives, hormone containing intrauterine device, depot injection, hormone implant, or sterilization (for contraception) plus condom (for prevention of reinfection). For male patients and partners of male patients who are of childbearing potential: use of two methods of effective contraception during the treatment period is mandatory (oral contraceptives, hormone containing intrauterine device, depot injection, hormone implant, or sterilization (for contraception) plus condom (for prevention of reinfection).

Exclusion Criteria:

For both subject groups (treatment arms 1 + 2):

1. Participation in an investigational trial within 30 days prior to enrollment and for the whole study duration.
2. Any current uncontrolled infection.
3. Current known acute or chronic infection with Hepatitis virus B or C.
4. Known Human immunodeficiency virus infection.
5. Subjects with known history of chronic (diabetes, hypertension, gastritis, etc.) or consuming diseases (cancer, multiple sclerosis, etc.), chronic inflammation, or liver or renal insufficiency.
6. Any chronic or acute condition including the skin, susceptible, in the opinion of the investigator, of interfering with the evaluation of the drug effect.
7. Laboratory data above the upper normal range.
8. Systemic intake of virostatics within 30 days prior to enrollment and for the whole study duration, with the exception of acyclovir and the related drugs famciclovir and valaciclovir.
9. Systemic intake of immunosuppressive or immuno-modulatory medication or vaccination within 30 days prior to enrollment and for the whole study duration.
10. Organ allograft recipient.
11. Medication intake, including over the counter products and dietary supplements such as iodine, fluoride, or vitamins, which would interfere with study results, except paracetamol and oral contraceptives, within one week before and during the study course. Subjects are not allowed to consume green, black or Oolong tea as well as red wine or any other beverages or foods containing green tea extract within three days before each blood sampling visit.
12. For female patients: pregnancy or lactation.
13. Blood transfusion within 30 days prior to enrollment.
14. Subjects who are placed in an institution due to a judicial or official directive.

    For patients (treatment arm 1, additionally):
15. Previous participation in a trial investigating sinecatechins in the treatment of external genital and perianal warts.
16. Treatment of external genital warts within 30 days prior to enrollment and for the whole study duration.
17. Current infection with Herpes genitalis or history of Herpes genitalis infection within the last 3 months prior to enrollment.
18. Any current and/or recurrent pathologically relevant genital infections other than genital warts.
19. Known allergies against any of the ingredients of the ointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of green tea catechins | Day 1/2 and Day 7/8
  Cmax, tmax, t1/2, AUC(0-t), and AUC of EGCg, EGC, ECg, and EC

CONTACTS AND LOCATIONS:
Overall Officials: Frank Wagner, Md, PD, Principal Investigator — Charité Research Organisation, Berlin
Locations (1):
- Charité Research Organisation, Berlin, Germany